CLINICAL TRIAL: NCT04096703
Title: Characterization of Lower Esophageal Sphincter Function in Idiopathic Esophagogastric Junction Outflow Obstruction and Clinical Response to Pneumatic Dilation
Brief Title: Idiopathic Esophagogastric Junction Outflow Obstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants for study.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00060689
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-11

CONDITIONS: Esophagogastric Junction Disorder
Keywords: Idiopathic Esophagogastric Junction Outflow Obstruction; Esophageal Sphincter Function; Esophagogastric Junction; Pneumatic Dilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Expectant management of EGJOO Group (No Intervention): The participants randomized to this group will receive expectant management of EGJOO. Expectant management is evaluating whether symptoms improve over time without an intervention
- Pneumatic dilation of EGJOO Group (Experimental): The participants randomized to the pneumatic dilation cohort will undergo an initial pneumatic dilation with a 30mm Rigiflex (Boston Scientific).
  Interventions: Procedure: Pneumatic dilation

INTERVENTIONS:
Procedure: Pneumatic dilation — The patients randomized to the pneumatic dilation cohort will undergo an initial pneumatic dilation with a 30mm Rigiflex (Boston Scientific). If the Eckardt score four weeks after initial dilation is > 4, then the patient will be scheduled for a second dilation with a 35mm Rigiflex balloon (Boston Scientific).
  Arms: Pneumatic dilation of EGJOO Group

SUMMARY:
This study compares two treatments for Idiopathic Esophagogastric Junction Outflow Obstruction: pneumatic dilation compared with expectant management, on symptoms and liquid barium emptying exams.

DETAILED DESCRIPTION:
The objectives of this study are to address these gaps in knowledge by:

Performing a randomized controlled trial in patients with idiopathic EGJOO that compares treatment outcomes after pneumatic dilation versus expectant management (disease controls) (expectant management). And, determining rational physiological and objective measures of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Initial HRIM consistent with the diagnosis of EGJOO and mechanical esophageal obstruction has been excluded by prior upper endoscopy.
* EGJOO patients with a retained liquid barium column on TBE ≥5cm in height at 1 minute
* Patients must have symptomatic dysphagia

Exclusion Criteria:

* Diseases that potentially could cause mechanical obstruction such as gastroesophageal reflux disease with erosive esophagitis, peptic stricture, cancer, eosinophilic esophagitis, prior fundoplication, adjustable gastric band surgery and hiatal hernias. Patients with any identifiable anatomic esophageal or gastric obstruction will be excluded from the study
* Patients with previous surgery on the esophagus or stomach
* Previous history of per oral endoscopic myotomy or prior pneumatic dilation
* History of gastroparesis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Brief esophageal dysphagia questionnaire (BEDQ) | Week 0
  The BEDQ is a 10-item self-report measure of dysphagia symptoms. The questionnaire is scored on a scale of 0-40. Higher scores indicate greater severity and frequency of dysphagia symptoms.
Brief esophageal dysphagia questionnaire (BEDQ) | 6 months
  The BEDQ is a 10-item self-report measure of dysphagia symptoms. The questionnaire is scored on a scale of 0-40. Higher scores indicate greater severity and frequency of dysphagia symptoms.
Eckardt Score | Week 0
  The Eckardt score is the grading system most frequently used for the evaluation of symptoms and efficacy of achalasia treatment. 33 It attributes points (0-3 points) to 4 symptoms of the disease (dysphagia, regurgitation, chest pain, and weight loss), and its total ranges from 0-12. The higher the score the worse the symptoms.
Eckardt Score | Week 4
  The Eckardt score is the grading system most frequently used for the evaluation of symptoms and efficacy of achalasia treatment. 33 It attributes points (0-3 points) to 4 symptoms of the disease (dysphagia, regurgitation, chest pain, and weight loss), and its total ranges from 0-12. The higher the score the worse the symptoms.
Eckardt Score | Week 6
  The Eckardt score is the grading system most frequently used for the evaluation of symptoms and efficacy of achalasia treatment. 33 It attributes points (0-3 points) to 4 symptoms of the disease (dysphagia, regurgitation, chest pain, and weight loss), and its total ranges from 0-12. The higher the score the worse the symptoms.
Number of participants with retained barium column ≥5cm | Week 6
  Measured in the timed barium esophagram

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clayton, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No